CLINICAL TRIAL: NCT04524247
Title: Impact of Frailty on Clinical Outcomes of Patients Treated for Thoracoabdominal and Complex Abdominal Aortic Aneurysms With Physician-Modified Fenestrated and Branched Stent Grafts
Brief Title: Frailty and Physician Modified Fenestrated Endograft for Thoracoabdominal Aortic Pathologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sukgu Han, MD, MS, Associate Professor of Surgery, Division of Vascular Surgery and Endovascular Therapy, University of Southern California, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-20-04282
Record Dates: First submitted 2020-08-15; First posted 2020-08-24 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Thoracoabdominal; Aortic, Aneurysm, Dissecting; Pararenal Aneurysm; Frailty Syndrome
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm; Frailty

STUDY DESIGN:
Intervention Model Description: Patients may be included in the study if the patient has at least one of the following indications and are anatomically appropriate for treatment with fenestrated/branched stent grafts.
  1. Pararenal, paravisceral, and type I to IV thoracoabdominal aortic aneurysms or chronic post-dissection aneurysms with a diameter 5cm or 2 times the normal aortic diameter.
  2. Aneurysm with a history of growth ≥ 0.5cm per year.
  3. Saccular aneurysms deemed at significant risk for rupture based on physician interpretation.
  4. Symptomatic aneurysm without hemodynamic instability
  5. Aneurysms meeting any of the above criteria 1~4, above or below the previous endovascular and/or open aortic repairs. Previously placed aortic stent graft or open aortic grafts may serve as seal zones.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PMEG FEVAR (Experimental): The only arm of this study will be enrolled subjects who undergo physician modified endografting as a treatment of their thoracoabdominal aortic aneurysms or complex abdominal aortic aneurysms.
  Interventions: Device: Physician Modified Endografts

INTERVENTIONS:
Device: Physician Modified Endografts — Modification procedure Description of modified device is detailed in Section 3.5 of IDE. In summary, the steps involved in modification of the Zenith Alpha thoracic stent grafts are;
  1. Unsheathing of the stent graft
  2. Retrieval of a trigger wire from the inner cannula of the delivery system
  3. Rerouting of the trigger wire along the stent graft
  4. Removal of proximal barbs.
  5. Creation of fenestrations and/or branch cuffs
  6. Placement of radiopaque markers around the fenestrations/ branch cuffs
  7. Placement of temporary and/or permanent diameter constraining ties
  8. (Optional) Placement of preloaded wires through the fenestrations/branch cuffs
  Other Names: Fenestrated, Branched Endografts

SUMMARY:
The primary objective of this single arm, prospective feasibility study, Impact of Frailty on Clinical Outcomes of Patients Treated for Thoracoabdominal and Complex Abdominal Aortic Aneurysms with Physician-Modified Fenestrated and Branched Stent Grafts, is to assess the use of the physician-modified fenestrated/branched endografts to repair thoracoabdominal and complex aortic aneurysms in subjects having appropriate anatomy, at high risks for open repairs. The primary intent of the study is to assess safety and preliminary effectiveness of the device acutely (i.e., treatment success and technical success), at 30 days (i.e., the rate of major adverse events (MAE)) and at 3 months, 6 months, 12 months, and annually to 5 years (i.e., the proportion of treatment group subjects that achieve and maintain treatment success).

Additionally, this study will assess the degree of patient frailty before and after the aneurysm repair, as well as the association between the preoperative baseline frailty and clinical outcomes detailed above. This will help improve subject selection in identification of high risk patients who would not only suffer poor clinical outcomes, but also experience decline in their functional status.

DETAILED DESCRIPTION:
Device Description

Two types of commercially approved thoracic aortic stent-grafts will be modified under the aegis of a physician-sponsored IDE protocol (G200159). The Cook (Bloomington, IN) Zenith Alpha proximal tapered mainbody thoracic stent-grafts and the Cook Zenith TX2 proximal tapered mainbody will be modified to form the fenestrated/branched aortic components. The Alpha thoracic stent-grafts are constructed of woven polyester graft sewn to discrete rows of self-expanding Nitinol Z stents. The most proximal sealing stent is located internally with fixation barbs that protrude through the graft material. The second proximal stent is straight, and the third stent is tapered by 4mm in diameter.

The diameter of the TX2 proximal tapered stent-grafts will range from 32mm to 42mm, depending on the size of the aorta at the proximal seal zone. The lengths will range from 154 to 210mm. The TX2 thoracic stent-grafts are constructed with woven polyester graft sewn to discrete rows of self-expanding stainless steel Z stents. The most proximal seal stent is sewn inside the polyester fabric. The third stent is tapered by either 4mm or 8mm in diameter.

The modification design will be planned using a 3-D multiplanar reconstruction analysis of the CT angiography. Proximal seal zone will be chosen at 2cm disease free parallel aortic walls. Target vessel position will be determined by the longitudinal distance between the proximal extent of the seal zone to the middle of the vessel orifice, as well as radial clock position. Based on these measurements, patient specific modification map will be constructed.

The modification will be designed to incorporate visceral and renal branches, utilizing a various combinations of fenestrations and branch cuffs. The choice between fenestrations and branch cuffs will be made based on the aortic size and angulation at the level of the target branches. For example, when the target branches are within the seal zone, fenestrations will be chosen. Conversely, branch cuffs will be incorporated onto the mainbody if the aorta at the level of the target branches is aneurysmal, or angulated where precise three dimensional position of the target branch, hence fenestration, along the implanted stent graft is difficult to predict.

Modification Technique

Modification will be performed on the day of the operation using strict sterile technique. Tapered low profile Cook Zenith Alpha proximal component thoracic stent grafts will be unsheathed. One of the trigger wires is retrieved from the inner cannula of the delivery system, to be used as a diameter constraining wire. This wire is rerouted posteriorly through and through the fabric of the stent graft using a long 22-gauge needle.

Fenestrations at planned locations will be created using an ophthalmic cautery, and reinforced with a double layer of Amplatz Gooseneck Snare (Medtronic, Minneapolis, MN) wires made up of braided Nitinol. The wires will be secured around the fenestration by tightly spaced 5-0 Ethibond (Ethicon, Somerville, NJ) locking sutures. Additional radiopaque markers will be sutured around each fenestration. When necessary, directional branch cuffs will be created by fashioning 8mm or 6mm Viabahn self expanding covered stents (Gore & Associates, Flagstaff, AZ) into 2cm long side branch cuffs. The branch cuffs will be sutured to the oval fenestration created on the aortic stent grafts by running 5-0 Goretex sutures. Radiopaque markers will be sutured around the entrance and exit of each branch cuff.

Prior to resheathing, the posterior aspect of Z-stents are constrained using loops of prolene sutures as diameter reducing ties. Proximal fixation barbs will be removed using a wire cutter. Fenestrations and branches designed to be catheterized from the brachial approach will be pre-wired with 0.014 inch guidewires. The modified stent graft will be resheathed using 2-0 Silk ties and Umbilical tapes.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be included in the study if the patient has at least one of the following indications and are anatomically appropriate for treatment with fenestrated/branched stent grafts.

  1. Pararenal, paravisceral, and type I to IV thoracoabdominal aortic aneurysms or chronic post-dissection aneurysms with a diameter 5cm or 2 times the normal aortic diameter.
  2. Aneurysm with a history of growth ≥ 0.5cm per year.
  3. Saccular aneurysms deemed at significant risk for rupture based on physician interpretation.
  4. Symptomatic aneurysm without hemodynamic instability
  5. Aneurysms meeting any of the above criteria 1~4, above or below the previous endovascular and/or open aortic repairs. Previously placed aortic stent graft or open aortic grafts may serve as seal zones.

Exclusion Criteria:

* Patients must be excluded from the study if any of the following conditions is true:

  1. Less than 18 years of age.
  2. Unwilling to comply with the follow-up schedule.
  3. Inability or refusal to give informed consent by the patient or a legally authorized representative.
  4. Pregnant or breastfeeding.
  5. Life-expectancy less than 2 years.
  6. Participation in another investigational clinical or device trial, with the exception of participation in another investigational endovascular stent-graft protocol and performed remotely from the fenestrated procedure (>30 days). Examples include remote (>30days) participation in a thoracic, or abdominal branch device trial.
  7. Eligible for treatment with FDA-approved marketed device.
  8. Eligible and willing to travel to a center with IDE protocol wherein the device is made by a manufacturer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2028-07-02 (Estimated); Study Completion 2032-07-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events | Immediately after the surgery up to 30 days. If the hospital stay exceeds 30 days, major adverse events that occur prior to discharge from hospital will be included.
  1. Aortic rupture within 30 days
  2. Lesion-related mortality within 30 days
  3. All-cause mortality within 30 days
  4. Permanent paraplegia, defined by lack of resolution at 1 month follow-up
  5. Permanent paraparesis, defined by lack of resolution at 1 month follow-up
  6. Renal function decline resulting in > 50% of estimated Glomerular Filtration Rate or New onset renal failure requiring dialysis, defined by ongoing dialysis at 1 month follow-up
  7. Severe bowel ischemia, requiring laparotomy
  8. Disabling stroke, reported within 30 days of the procedure, without resolution at 90 days post-procedure
  9. Myocardial infarction
  10. Respiratory failure requiring prolonged (> 24 hours from anticipated) mechanical ventilation or reintubation

SECONDARY OUTCOMES:
Rate of Technical Success | Immediately after the surgery
  Successful delivery of the device(s) to the intended target implantation site(s), and successful removal of the delivery system
Rate of Treatment Success | 30-days, 6 months, 12 months, 18 months, 2 years, 3 years, 4 years, 5 years
  Treatment Success is defined by having met ALL of the following dichotomous conditions.
  * Technical success (Yes/No)
  * Absence of death form the initial procedure, secondary intervention for aortic-related cause (Yes/No)
  * Absence of persistent type I or III endoleaks (Yes/No)
  * Absence of aneurysm sac expansion > 5mm (Yes/No)
  * Absence of device migration > 10mm (Yes/No)
  * Absence of failure due to device integrity issues (Yes/No)
  * Absence of aneurysm rupture (Yes/No)
  * Absence of conversion to open surgical repair (Yes/No)
  * Absence of permanent paraplegia, disabling stroke, or dialysis that resulted from the initial operation or a secondary intervention to treat the original aortic pathology (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Sukgu M Han, MD, MS, Principal Investigator — University of Southern California
Locations (1):
- Keck Hospital of University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uflacker R, Robison JD, Schonholz C, Ivancev K. Clinical experience with a customized fenestrated endograft for juxtarenal abdominal aortic aneurysm repair. J Vasc Interv Radiol. 2006 Dec;17(12):1935-42. doi: 10.1097/01.RVI.0000248828.92093.1A. PMID 17185689
- [Background] Amiot S, Haulon S, Becquemin JP, Magnan PE, Lermusiaux P, Goueffic Y, Jean-Baptiste E, Cochennec F, Favre JP; Association Universitaire de Recherche en Chirurgie Vasculaire. Fenestrated endovascular grafting: the French multicentre experience. Eur J Vasc Endovasc Surg. 2010 May;39(5):537-44. doi: 10.1016/j.ejvs.2009.12.008. Epub 2010 Jan 25. PMID 20093051
- [Background] Verhoeven EL, Katsargyris A, Bekkema F, Oikonomou K, Zeebregts CJ, Ritter W, Tielliu IF. Editor's Choice - Ten-year Experience with Endovascular Repair of Thoracoabdominal Aortic Aneurysms: Results from 166 Consecutive Patients. Eur J Vasc Endovasc Surg. 2015 May;49(5):524-31. doi: 10.1016/j.ejvs.2014.11.018. Epub 2015 Jan 17. PMID 25599593
- [Background] Mastracci TM, Greenberg RK, Eagleton MJ, Hernandez AV. Durability of branches in branched and fenestrated endografts. J Vasc Surg. 2013 Apr;57(4):926-33; discussion 933. doi: 10.1016/j.jvs.2012.09.071. Epub 2013 Feb 20. PMID 23433817
- [Background] O'Neill S, Greenberg RK, Haddad F, Resch T, Sereika J, Katz E. A prospective analysis of fenestrated endovascular grafting: intermediate-term outcomes. Eur J Vasc Endovasc Surg. 2006 Aug;32(2):115-23. doi: 10.1016/j.ejvs.2006.01.015. Epub 2006 Mar 31. PMID 16580236
- [Background] British Society for Endovascular Therapy and the Global Collaborators on Advanced Stent-Graft Techniques for Aneurysm Repair (GLOBALSTAR) Registry. Early results of fenestrated endovascular repair of juxtarenal aortic aneurysms in the United Kingdom. Circulation. 2012 Jun 5;125(22):2707-15. doi: 10.1161/CIRCULATIONAHA.111.070334. PMID 22665884
- [Background] Reilly LM, Rapp JH, Grenon SM, Hiramoto JS, Sobel J, Chuter TA. Efficacy and durability of endovascular thoracoabdominal aortic aneurysm repair using the caudally directed cuff technique. J Vasc Surg. 2012 Jul;56(1):53-63; discussion 63-4. doi: 10.1016/j.jvs.2012.01.006. Epub 2012 May 3. PMID 22560233
- [Background] Starnes BW, Heneghan RE, Tatum B. Midterm results from a physician-sponsored investigational device exemption clinical trial evaluating physician-modified endovascular grafts for the treatment of juxtarenal aortic aneurysms. J Vasc Surg. 2017 Feb;65(2):294-302. doi: 10.1016/j.jvs.2016.07.123. Epub 2016 Sep 26. PMID 27687323
- [Background] Scali ST, Neal D, Sollanek V, Martin T, Sablik J, Huber TS, Beck AW. Outcomes of surgeon-modified fenestrated-branched endograft repair for acute aortic pathology. J Vasc Surg. 2015 Nov;62(5):1148-59.e2. doi: 10.1016/j.jvs.2015.06.133. Epub 2015 Aug 5. PMID 26254453
- [Background] Tsilimparis N, Heidemann F, Rohlffs F, Diener H, Wipper S, Debus ES, Kolbel T. Outcome of Surgeon-Modified Fenestrated/Branched Stent-Grafts for Symptomatic Complex Aortic Pathologies or Contained Rupture. J Endovasc Ther. 2017 Dec;24(6):825-832. doi: 10.1177/1526602817729673. Epub 2017 Sep 6. PMID 28874089
- [Background] Georgiadis GS, van Herwaarden JA, Antoniou GA, Hazenberg CE, Giannoukas AD, Lazarides MK, Moll FL. Systematic Review of Off-the-Shelf or Physician-Modified Fenestrated and Branched Endografts. J Endovasc Ther. 2016 Feb;23(1):98-109. doi: 10.1177/1526602815611887. Epub 2015 Oct 23. PMID 26496957
- [Background] O'Donnell TFX, Patel VI, Deery SE, Li C, Swerdlow NJ, Liang P, Beck AW, Schermerhorn ML. The state of complex endovascular abdominal aortic aneurysm repairs in the Vascular Quality Initiative. J Vasc Surg. 2019 Aug;70(2):369-380. doi: 10.1016/j.jvs.2018.11.021. Epub 2019 Feb 2. PMID 30718110
- [Background] Han SM, Tenorio ER, Mirza AK, Zhang L, Weiss S, Oderich GS. Low-profile Zenith Alpha Thoracic Stent Graft Modification Using Preloaded Wires for Urgent Repair of Thoracoabdominal and Pararenal Abdominal Aortic Aneurysms. Ann Vasc Surg. 2020 Aug;67:14-25. doi: 10.1016/j.avsg.2020.02.022. Epub 2020 Mar 20. PMID 32205248